CLINICAL TRIAL: NCT02781415
Title: Comparison of Acupuncture and Titrated (TM) Morphine in Patients Presenting to the Emergency Room (ER) With Acute Renal Colic (RC)
Brief Title: Acupuncture Versus Titrated Morphine in Patients With Renal Colic
Acronym: AcuRC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Clinical Professor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14/25
Record Dates: First submitted 2016-05-16; First posted 2016-05-24 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Renal Colic
MeSH Terms: conditions — Renal Colic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture (Experimental): Traditional Acupuncture Session:Patients in this group will benefit from a 30 minutes acupuncture session made by an experimented physician.
  Interventions: Procedure: Traditional Acupuncture Session
- Titrated Morphine (Active Comparator): Morphine Titration:Patients will receive an intravenous titration of morphine by a qualified nurse.
  Interventions: Drug: Morphine Titration

INTERVENTIONS:
Procedure: Traditional Acupuncture Session — Skin disinfection was made by an antiseptic solution in the sites of insertion and sterile acupuncture needles were used (0.25 x 0.5 mm).
  Patients were installed in a seated position and needles were inserted perpendicularly through the skin to a depth of 1 - 2 cm until the "De Qi" was achieved.
  The "DeQi" corresponds to a feeling of numbness and tingling within the range of acupoint, The insertion sites are represented by the urinary bladder meridian points to the side of the pain (UB21, UB22, UB23, UB24, UB26, UB45, UB46, UB47, UB48 and UB49).
  Arms: Acupuncture
Drug: Morphine Titration — Morphine was previously prepared by a study nurse by diluting a 10 mg / 1 ml flakon of morphine chlorhydrate in a 9 ml solution of serum saline to obtain a 10 ml preparation (1 ml = 1 mg).
  An initial bolus of 0.1 mg per Kg of actual body weight of morphine chlorhydrate solution is administered.
  A titration dose of 0.1 mg / Kg of body weight was repeated every 5 minutes' interval until reaching the therapeutic goal.
  Arms: Titrated Morphine

SUMMARY:
The aim of this study is to compare the clinical efficacy and safety profiles of a 30 minutes acupuncture session performed at an ER of a tertiary hospital versus titrated intravenous morphine in the management of acute severe pain syndromes (defined as a visual analogue scale (VAS) score >/= 70) taking for example acute renal colic.

DETAILED DESCRIPTION:
acupuncture session performed at an ER of a tertiary hospital versus titrated intravenous morphine in the management of acute severe pain syndromes (defined as a visual analogue scale (VAS) score >/= 70) taking for example acute renal colic.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* Presenting with acute non complicated renal colic
* Baseline VAS score >/= 70

Exclusion Criteria:

* complicated renal colic
* VAS score < 70
* Pain of traumatic origin
* Coagulation abnormalities
* Skin affections impairing the use of pre-specified insertion points
* Enable to use the VAS
* Patients who received analgesics less than 6 hours prior to enrollment
* Patients refusing or enable to give written informed consent
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Pain score Change | at baseline and 10, 20, 30, 45 and 60 minutes after the start of intervention
  Pain score is measured by a 100 millimeter visual analogue scale (VAS) and corresponds to the severity of the pain felt by the patient and varying from 0 (corresponding to no pain) to 100 (corresponding to the maximum imaginable pain).

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | during the 1 hour protocol and up to 2 hours after
  Corresponds to the occurence of side effects related to the intervention. Side effects occurence is evaluated via a checklist for each study group and the degree of amputability is evaluated via a 3 point likert scale (1: not probable, 2: probable and 3 : very probable / almost certain).
  In the morphine group we followed patients for the occurence of drowsiness, dizziness, nausea and vomiting, respiratory distress and hypotension.
  In the acupuncture group we followed patients for the occurence of local rush / bleeding / itching, needle blockage and fainting

CONTACTS AND LOCATIONS:
Overall Officials: Nouira Semir, Professor, Principal Investigator — University Hospital of Monastir
Locations (1):
- Fattouma Bourguiba University Hospital, Monastir, Monastir Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: Yes